CLINICAL TRIAL: NCT06165536
Title: Laryngeal and Vocal Tract Strategies to Reduce Vocal Fold Contact Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Zhaoyan Zhang, PhD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-001058; R01DC020240 (NIH)
Record Dates: First submitted 2023-11-27; First posted 2023-12-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Mid-membranous Vocal Fold Lesion
Keywords: Vocal fold lesion; Vocal hyperfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voice therapy (Other): Resonant voice therapy is a standard of care procedure for treating phonotraumatic vocal hyperfunction. The full standardized voice therapy program will have a duration of four weeks, each week with one 60-minute therapy session.
  Interventions: Behavioral: Resonant voice therapy

INTERVENTIONS:
Behavioral: Resonant voice therapy — Resonant voice therapy is a standard of care procedure for treating phonotraumatic vocal hyperfunction. The full standardized voice therapy program will have a duration of four weeks, each week with one 60-minute therapy session.

SUMMARY:
Phonotraumatic vocal hyperfunction is one of the most frequently occurring conditions to affect the voice. This voice disorder often involves vocal fold injury due to repeated, excessive contact pressure between the vocal folds when they collide during voice production. In the clinic, voice therapy attempts to modify unhealthy vocal behaviors through different techniques or exercises. While voice therapy is generally considered effective, the scientific rationale for its therapeutic benefits still remains unclear. It is generally believed that these exercises lead to adjustments in the larynx and vocal tract that reduce vocal fold contact pressure. However, this assumption has never been tested in humans or laboratory experiments. The goal of this clinical trial is to investigate the effectiveness of voice therapy in reducing vocal fold contact pressures and in eliciting the hypothesized favorable laryngeal and vocal tract configurations.

DETAILED DESCRIPTION:
This study will investigate the degree to which a well-documented voice therapy technique, resonant voice therapy, reduces vocal fold contact pressure compared to baseline, and which if any laryngeal and vocal tract adjustments occur in association with this phonation pattern. The investigators will measure contact pressure in vivo in human subjects, and will use computed tomography scans to assess laryngeal and vocal tract configurations before and after initial voice training, in adults with phonotraumatic lesions. The investigators will correlate these measures to patient-reported outcome measures and other secondary outcome measures across longer-term therapy. It is hypothesized that findings regarding favorable physical adjustments associated with reduction in contact pressure shown in this aim will match those identified in our recent simulation studies, and that initial reduction in contact pressure in resonant voice, associated with relevant perceptual, acoustic, and subglottic pressure changes, will correlate with improved long-term voice therapy outcome.

Patients will be those who have been diagnosed by a fellowship trained laryngologist with bilateral mid-membranous lesions that by appearance and history are phonotraumatic and who are referred to resonant voice therapy (RVT). Each subject will receive resonant voice therapy, a standard of care procedure for treating phonotraumatic vocal hyperfunction. The full standardized voice therapy program will have a duration of four weeks, each week with one 60-minute therapy session. All voice therapy sessions will be video recorded. Ten percent of recordings will be randomly selected and used in fidelity checks. Data collection will take place at 3 time points: before therapy (baseline), immediately after an initial therapy session, and after 4 weeks of therapy. At baseline, each subject will fill out a Voice Handicap Index-10 (VHI-10) questionnaire, and will receive videoendoscopic examination, CT scans of the head and neck region during phonation, acoustic and subglottal pressure measurement, and contact pressure measurement. Data collection will be repeated the same day following an initial session of RVT training. Same-day data collection will ensure that lesion characteristics have not changed from baseline, and avoid confounding effects of lesion change in contact pressure measures. Degree of resonant voice acquisition will be determined by speech language pathologists (SLPs) real-time and will be further characterized quantitatively by post hoc perceptual evaluation and acoustic measures. Finally, after 4 weeks of RVT, follow-up measure will include VHI-10, endoscopic exam, perceptual, acoustic, and subglottal pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40 years (to minimize developmental changes associated with adolescent and elderly age)
* Clinic diagnosis by a fellowship trained laryngologist of mid-membranous lesions that by history and appearance are phonotraumatic
* Must be referred for voice therapy

Exclusion Criteria:

* Medical comorbidities (e.g., autoimmune disorders) beyond seasonal allergy and laryngopharyngeal reflux
* Vocal fold lesions generally regarded to be less responsive to voice therapy (e.g. vocal fold cysts).
* Claustrophobia
* Inability to replicate fundamental frequencies required for the study at the intensity levels determined

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Voice handicap index (VHI-10) | 30 minutes before the first voice therapy session, and 30 minutes after the last session of the 4-week voice therapy
  VHI-10 scores will be measured using the voice handicap index-10 questionnaire. Scores for the VHI-10 range from 0 to 40, with higher scores indicating a greater voice-related handicap.
Severity of vocal fold lesions | 30 minutes before the first voice therapy session, and 30 minutes after the last session of the 4-week voice therapy
  The medical severity of vocal fold lesions will be rated based on videoendoscopic examination of the larynx. The Nuss scale - a vetted, widely clinically used visual-perceptual scale - will be used to rate presence/absence of nodules (0) and nodules size (1 = small, 2 = moderate, 3 = large). Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Perceptual evaluation of voice | Perceptual evaluation will be performed within 6 months of data collection, using voices recorded 30 minutes before and 30 minutes after the first voice therapy session and 30 minutes after the last session of the 4-week voice therapy
  Perceptual evaluation will be conducted on the recorded phrase, "We were away a year ago," using the Overall Severity scale from the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V), using pre-post therapy paired comparison procedures. Scores will range between 0 and 100, with higher scores indicating worse outcomes. Raters will be five blinded voice-specialized speech language pathologists otherwise not involved with the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyan Zhang, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Rehab Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected during this project, including acoustic, aerodynamic, vocal fold geometry data from medial surface imaging or CT scans, vocal fold contact pressure, will be archived and made available to interested investigators on request after the investigators have finished planned analyses and publications.
Supporting Information: Study Protocol, SAP
Time Frame: After the investigators have finished planned analyses and publications
Access Criteria: Data will be made available to interested investigators upon request to and reviewed by the principal investigator.